CLINICAL TRIAL: NCT06660680
Title: The Ethics Committee of the Second Hospital of Chinese Medicine
Brief Title: The Effect of Methylene Blue Infiltrating Injection on Anal Pain After Milligan-Morgan Surgery: a Randomized Controlled Clinical Study
Acronym: MBI
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Heng Deng, the second Hospital of Chinese Medicine, The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFBH2021011; (No. 2023AH050848) (Other Grant/Funding Number: Scientific Research Project of Colleges and Universities of Anhui Province)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Mixed Hemorrhoids
Keywords: Milligan-Morgan surgery
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): received MBI treatment to their surgical incisions upon completion of surgery
  Interventions: Drug: Methylene Blue
- Control group (No Intervention): administered lornoxicam on an as-needed basis for analgesia.

INTERVENTIONS:
Drug: Methylene Blue — Received MBI treatment to their surgical incisions upon completion of surgery
  Arms: Study Group

SUMMARY:
A variety of analgesic strategies are available following mixed hemorrhoids surgery, including pharmacological interventions (7), acupuncture, moxibustion, and electroacupuncture . Medications such as opioid analgesics and non-steroidal anti-inflammatory drugs (NSAIDs) are commonly used but can be associated with side effects including nausea, vomiting, and gastrointestinal bleeding, with long-term use potentially leading to addiction (8). Complementary therapies require skilled administration and regular treatment sessions.

Methylene blue (MB), a cationic thiazine dye extensively utilized as a biological stain and chemical indicator, has been increasingly recognized for its potential analgesic properties (9). In the present study, methylene blue infiltrating injection (MBI) was administered to treat anal pain resulting from Milligan-Morgan surgery, with the aim of assessing its analgesic efficacy and safety profile.

ELIGIBILITY:
Inclusion Criteria:①Alignment with the diagnostic criteria for mixed hemorrhoids as outlined in the "American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Hemorrhoids" ; ②Provision of informed consent following a thorough comprehension of the study's aims; ③An age bracket of 18 to 75 years; ④Satisfaction of surgical indications.

-

Exclusion Criteria:①Presence of anal fistula, anal fissure, perianal abscess, enteritis, or other intestinal pathologies; ②Patients with known allergies; ③Impaired liver or kidney function; ④Pregnancy or lactation.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain | pain scores at 6, 24, 48, and 72 hours postoperatively
  Visual Analog Scale (VAS) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Second hospital affiliated Anhui University of Chinese Medicine, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anorectal Branch of Chinese Medical Doctor A, Colorectal Surgery Group SSoCMA.